CLINICAL TRIAL: NCT00613457
Title: AIEOP LLA 2000 Multicenter Study for the Diagnosis and Treatment of Childhood Acute Lymphoblastic Leukemia
Brief Title: Combination Chemotherapy Based on Risk of Relapse in Treating Young Patients With Acute Lymphoblastic Leukemia
Acronym: AIEOP LLA 2000
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Associazione Italiana Ematologia Oncologia Pediatrica (Other)
Responsible Party: Giuseppe Masera MD, Clinica Pediatrica Università di MIlano Bicocca
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AIEOP LLA 2000; AIEOP LLA 2000
Record Dates: First submitted 2008-01-21; First posted 2008-02-13 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Leukemia
MeSH Terms: conditions — Leukemia | interventions — Dexamethasone; Asparaginase; Cyclophosphamide; Cytarabine; Daunorubicin; Doxorubicin; Etoposide; Ifosfamide; Mercaptopurine; Methotrexate; Prednisone; Thioguanine; Vincristine; Vindesine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- I (Experimental): o Arm I (closed to accrual as of 6/30/2006): Patients receive prednisone (PRED) on days 8-28.
  Interventions: Drug: asparaginase; Drug: cyclophosphamide; Drug: cytarabine; Drug: daunorubicin; Drug: mercaptopurine; Drug: Methotrexate; Drug: prednisone; Drug: Vincristine
- II (Experimental): o Arm II (closed to accrual as of 6/30/2006): Patients receive dexamethasone (DEXA) on days 8-28.
  Interventions: Drug: dexamethasone; Drug: asparaginase; Drug: cyclophosphamide; Drug: cytarabine; Drug: daunorubicin; Drug: mercaptopurine; Drug: Methotrexate; Drug: Vincristine
- Reintensification Arm I (Experimental): o Arm I (standard reinduction therapy, protocol II [closed to accrual as of 6/30/2006]): SR and IR patients receive DEXA on days 1-22; VCR and doxorubicin hydrochloride (DOX) in weeks 2-5; ASP on days 8, 11, 15, and 18; CPM on day 36; ARA-C and thioguanine (TG) on days 36-49; and MTX IT on days 38 and 45. Patients then proceed to maintenance therapy.
  Interventions: Drug: Asparaginase; Drug: cyclophosphamide; Drug: cytarabine; Drug: doxorubicin; Drug: mercaptopurine; Drug: Methotrexate; Drug: thioguanine; Drug: Vincristine
- Reintensification Arm II (Experimental): • Arm II (reduced-intensity reinduction therapy, protocol III [closed to accrual as of 6/30/2006]): SR patients receive DEXA on days 1-15; VCR and DOX on days 1 and 8; ASP on days 1, 4, 8, and 11; CPM on day 15; ARA-C and TG on days 15-28; and MTX IT on days 16 and 23. Patients then proceed to maintenance therapy.
  Interventions: Drug: Asparaginase; Drug: cyclophosphamide; Drug: cytarabine; Drug: doxorubicin; Drug: mercaptopurine; Drug: Methotrexate; Drug: thioguanine; Drug: Vincristine
- Reintensification Arm III (Experimental): • Arm III (reduced-intensity reinduction/second delayed reinduction therapy [double reintensification therapy] [closed to accrual as of 6/30/2006]): IR patients receive reduced-intensity reintensification therapy as in arm II. After a 10-week interim maintenance phase, treatment repeats once for a second delayed course of reintensification therapy. Patients then proceed to maintenance therapy.
  Interventions: Drug: Asparaginase; Drug: cytarabine; Drug: doxorubicin; Drug: mercaptopurine; Drug: Methotrexate; Drug: Vincristine
- Reintensification Arm IV (Experimental): • Arm IV (standard reintensification therapy [closed to accrual as of 6/30/2006]): HR patients receive one sequence of the following HR therapy elements, in this order: 1, 2, 3, following standard reinduction therapy protocol II repeated twice after a four weeks Interim Maintenance phase. Patients then proceed to maintenance therapy.
  * Element HR-1: Patients receive DEXA on days 1-5; VCR on days 1 and 6; ARA-C twice on day 5; MTX and CPM every 12 hours on days 2-4 (5 doses); ASP on day 6 ; and MTX/ARA-C/PRED IT on day 1.
  * Element HR-2: Patients receive DEXA on days 1-5; vindesine on days 1 and 6; DNR on day 5; MTX and ifosfamide every 12 hours on days 2-4 (5 doses); ASP on day 6; and MTX/ARA-C/PRED IT on day 1.
  * Element HR-3: Patients receive DEXA on days 1-5; ARA-C every 12 hours on days 1-2 (4 doses); etoposide five times daily on days 3-5; ASP on day 5; and MTX/ARA-C/PRED IT on day 1.
  Interventions: Drug: Etoposide; Drug: Ifosfamide; Drug: Methotrexate; Drug: Vincristine; Drug: Vindesine
- Reintensification Arm V (Experimental): • Arm V (extended reintensification therapy [triple protocol III] [closed to accrual as of 6/30/2006]): HR patients receive HR therapy elements 3, 2, and 1 following reintensification therapy repeated the therapy element three times with 4-week interim maintenance phases in between. Patients then proceed to maintenance therapy.
  * Interim maintenance/maintenance therapy: Patients receive MTX once weekly and MP daily until week 104 plus IT MTX every eight weeks.
  * Radiotherapy: HR patients or patients with T-cell acute lymphoblastic leukemia or CNS disease undergo CNS radiotherapy.
  Interventions: Drug: Etoposide; Drug: Ifosfamide; Drug: Methotrexate; Drug: Vincristine; Drug: Vindesine

INTERVENTIONS:
Drug: dexamethasone — 10 mg/sqm/day from for 21 days
  Arms: II
Drug: asparaginase — native E-coli Asparaginase 5,000 IU/sqm x 8 doses
  Arms: I; II
Drug: Asparaginase — native E-Coli Asparaginase 10,000 IU/sqm x 4 doses
  Arms: Reintensification Arm I; Reintensification Arm II; Reintensification Arm III
Drug: cyclophosphamide — 1,000 mg/sqm i.v. 2 doses in Induction phase 1000 mg/sqm i.v. 1 dose in Protocoll II 500 mg/sqm i.v. 1 dose in protocol III
  Arms: I; II; Reintensification Arm I; Reintensification Arm II
Drug: cytarabine — 75 mg/sqm i.v.or s.c. 4 doses/week for 4 weeks in Induction phase 75 mg/sqm i.v.or s.c. 4 doses/week for 2 weeks in Protocol II and III
  Arms: I; II; Reintensification Arm I; Reintensification Arm II; Reintensification Arm III
Drug: daunorubicin — 30 mg/sqm i.v. 4 doses in Induction phase
  Arms: I; II
Drug: doxorubicin — 30 mg/sqm i.v. x 4 doses in Protocol II and III
  Arms: Reintensification Arm I; Reintensification Arm II; Reintensification Arm III
Drug: Etoposide — 100 mg/sqm i.v. for 3 doses in HR block 3
  Arms: Reintensification Arm IV; Reintensification Arm V
Drug: Ifosfamide — 800 mg/sqm i.v.q12h x 5 in HR block 2
  Arms: Reintensification Arm IV; Reintensification Arm V
Drug: mercaptopurine — 60 mg/sqm p.o. c 28 days in Induction phase 60 mg/sqm p.o. x 56 days in Protocol M 50 mg/sqm daily in Maintenance phase
  Arms: I; II; Reintensification Arm I; Reintensification Arm II; Reintensification Arm III
Drug: Methotrexate — by age i.t. in Induction/Protocol M/Protocol II/Protocol III/HR Blocks and maintenance
Drug: prednisone — 60 mg/sqm daily p.o. for 28 days then tapered in Induction phase
  Arms: I
Drug: thioguanine — 60 mg/sqm p.o. x 14 days in Protocol II and Protocol III
  Arms: Reintensification Arm I; Reintensification Arm II
Drug: Vincristine — 1.5 mg/sqm i.v. x 4 doses in Induction phase and Protocol II 1.5 mg/sqm i.v. x 2 doses in Protocol III and HR block 1
Drug: Vindesine — 3 mg/sqm i.v. x 2 doses in HR block 2
  Arms: Reintensification Arm IV; Reintensification Arm V

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more cancer cells. It is not yet known which combination chemotherapy regimen is more effective in treating young patients with acute lymphoblastic leukemia.

PURPOSE: Thisphase III trial is studying several different combination chemotherapy regimens to compare how well they work in treating young patients with acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the relative efficacy of induction therapy comprising dexamethasone or prednisone, in terms of a higher rate of event-free survival (EFS) and overall survival and a reduced rate of relapse, in pediatric patients with intermediate-risk or high-risk acute lymphoblastic leukemia (ALL).
* Compare the relative safety of a reduced-intensity reintensification regimen comprising dexamethasone, vincristine, cyclophosphamide, and anthracyclines vs a standard treatment regimen in pediatric patients with standard-risk ALL identified by fast clearance of leukemic cells.
* Compare the efficacy of a second delayed reintensification regimen vs standard reintensification therapy, in terms of improved EFS, in pediatric patients with intermediate-risk ALL.
* Compare the efficacy of extended reintensification therapy (triple reinduction) vs standard reintensification therapy (intensive pulses and one reintensification) in pediatric patients with high-risk ALL.

OUTLINE: This is a randomized, multicenter study.

* Prednisone prephase therapy: Patients receive oral prednisone on days 1-7 and one dose of methotrexate (MTX) intrathecally (IT) on day 1.
* Induction/consolidation therapy, protocol I: Patients are randomized to 1 of 2 treatment arms.

  * Arm I (closed to accrual as of 6/30/2006): Patients receive prednisone (PRED) on days 8-28.
  * Arm II (closed to accrual as of 6/30/2006): Patients receive dexamethasone (DEXA) on days 8-28.

Patients in both arms also receive vincristine (VCR) and daunorubicin hydrochloride (DNR) once weekly in weeks 2-5; asparaginase (ASP) on days 12-33; cyclophosphamide (CPM) on days 36 and 64; cytarabine (ARA-C) in weeks 6-9; mercaptopurine (MP) on days 36-63; and MTX IT on days 1, 15, 29,38 and 52.* NOTE: *Patients with CNS disease also receive MTX IT on days 8 and 22. After completion of induction/consolidation therapy, patients are stratified according to risk group based on disease response (standard-risk [SR] group [negative minimal residual disease (MRD) on day 33 and before protocol M, day 78] vs high-risk [HR] group [MRD ≥ 10^-³ on day 78] vs intermediate-risk [IR] group [all nonSR/nonHR]).* Patients with SR and IR disease proceed to consolidation therapy-protocol M. Patients with HR disease proceed to HR block therapy.

NOTE: *Patients meeting any of the following criteria are placed in the HR group regardless of MRD response: Philadelphia chromosome-positive disease (BCR/ABL or t[9;22]; translocations [t4;11][q11;q23] or MLL/AF4); "prednisone-poor-response" (≥ 1,000 blasts/mm³ in the peripheral blood on day 8 after prednisone prephase therapy); or no response to study induction therapy (M2/3 at day 33).

• Consolidation, protocol M: Patients receive MP on days 1-56 and MTX on days 8, 22, 36, and 50.

After completion of extracompartment therapy, SR and IR patients proceed to reintensification therapy. SR patients are randomized to arms I or II. IR patients are randomized to arms I or III. HR patients who have completed induction/consolidation therapy are randomized to arms IV or V.

* Reinduction therapy:

  o Arm I (standard reinduction therapy, protocol II [closed to accrual as of 6/30/2006]): SR and IR patients receive DEXA on days 1-22; VCR and doxorubicin hydrochloride (DOX) in weeks 2-5; ASP on days 8, 11, 15, and 18; CPM on day 36; ARA-C and thioguanine (TG) on days 36-49; and MTX IT on days 38 and 45. Patients then proceed to maintenance therapy.
* Arm II (reduced-intensity reinduction therapy, protocol III [closed to accrual as of 6/30/2006]): SR patients receive DEXA on days 1-15; VCR and DOX on days 1 and 8; ASP on days 1, 4, 8, and 11; CPM on day 15; ARA-C and TG on days 15-28; and MTX IT on days 16 and 23. Patients then proceed to maintenance therapy.
* Arm III (reduced-intensity reinduction/second delayed reinduction therapy [double reintensification therapy] [closed to accrual as of 6/30/2006]): IR patients receive reduced-intensity reintensification therapy as in arm II. After a 10-week interim maintenance phase, treatment repeats once for a second delayed course of reintensification therapy. Patients then proceed to maintenance therapy.
* Arm IV (standard reintensification therapy [closed to accrual as of 6/30/2006]): HR patients receive one sequence of the following HR therapy elements, in this order: 1, 2, 3, following standard reinduction therapy protocol II repeated twice after a four weeks Interim Maintenance phase. Patients then proceed to maintenance therapy.

  * Element HR-1: Patients receive DEXA on days 1-5; VCR on days 1 and 6; ARA-C twice on day 5; MTX and CPM every 12 hours on days 2-4 (5 doses); ASP on day 6 ; and MTX/ARA-C/PRED IT on day 1.
  * Element HR-2: Patients receive DEXA on days 1-5; vindesine on days 1 and 6; DNR on day 5; MTX and ifosfamide every 12 hours on days 2-4 (5 doses); ASP on day 6; and MTX/ARA-C/PRED IT on day 1.
  * Element HR-3: Patients receive DEXA on days 1-5; ARA-C every 12 hours on days 1-2 (4 doses); etoposide five times daily on days 3-5; ASP on day 5; and MTX/ARA-C/PRED IT on day 1.
* Arm V (extended reintensification therapy [triple protocol III] [closed to accrual as of 6/30/2006]): HR patients receive HR therapy elements 3, 2, and 1 following reintensification therapy repeated the therapy element three times with 4-week interim maintenance phases in between. Patients then proceed to maintenance therapy.

  * Interim maintenance/maintenance therapy: Patients receive MTX once weekly and MP daily until week 104 plus IT MTX every eight weeks.
  * Radiotherapy: HR patients or patients with T-cell acute lymphoblastic leukemia or CNS disease undergo CNS radiotherapy.

PROJECTED ACCRUAL: A total of 2,039 patients has been accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed acute lymphoblastic leukemia (ALL)
* No secondary ALL
* More than 4 weeks since prior chemotherapy
* More than 4 weeks since prior steroids

Exclusion Criteria:

* Prior disease that would preclude treatment with chemotherapy

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2039 (Actual)
Dates: Start 2000-09; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Efficacy of dexamethasone vs prednisone during the induction phase | 5 years
Event-free survival (EFS) and overall survival after initial remission in intermediate-risk and high-risk patients | 5 years
Safety and efficacy of treatment reduction during reintensification in standard-risk patients | 5 years
EFS after second delayed reintensification in intermediate-risk patients | 5 years
Outcome after extended reintensification therapy in high-risk patients | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Masera, MD, Study Chair — Clinica Pediatrica Università di milano Bicocca

REFERENCES:
- [Derived] Heilmann J, Vieth S, Moricke A, Attarbaschi A, Barbaric D, Bodmer N, Colombini A, Dalla-Pozza L, Elitzur S, Izraeli S, Mann G, Niggli F, Silvestri D, Stary J, Rizzari C, Valsecchi MG, Zapotocka E, Zimmermann M, Cario G, Schrappe M, Conter V. Effect of two additional doses of intrathecal methotrexate during induction therapy on serious infectious toxicity in pediatric patients with acute lymphoblastic leukemia. Haematologica. 2023 Dec 1;108(12):3278-3286. doi: 10.3324/haematol.2022.281788. PMID 37021527
- [Derived] Cario G, Leoni V, Conter V, Attarbaschi A, Zaliova M, Sramkova L, Cazzaniga G, Fazio G, Sutton R, Elitzur S, Izraeli S, Lauten M, Locatelli F, Basso G, Buldini B, Bergmann AK, Lentes J, Steinemann D, Gohring G, Schlegelberger B, Haas OA, Schewe D, Buchmann S, Moericke A, White D, Revesz T, Stanulla M, Mann G, Bodmer N, Arad-Cohen N, Zuna J, Valsecchi MG, Zimmermann M, Schrappe M, Biondi A. Relapses and treatment-related events contributed equally to poor prognosis in children with ABL-class fusion positive B-cell acute lymphoblastic leukemia treated according to AIEOP-BFM protocols. Haematologica. 2020 Jul;105(7):1887-1894. doi: 10.3324/haematol.2019.231720. Epub 2019 Oct 10. PMID 31601692
- [Derived] Schrappe M, Bleckmann K, Zimmermann M, Biondi A, Moricke A, Locatelli F, Cario G, Rizzari C, Attarbaschi A, Valsecchi MG, Bartram CR, Barisone E, Niggli F, Niemeyer C, Testi AM, Mann G, Ziino O, Schafer B, Panzer-Grumayer R, Beier R, Parasole R, Gohring G, Ludwig WD, Casale F, Schlegel PG, Basso G, Conter V. Reduced-Intensity Delayed Intensification in Standard-Risk Pediatric Acute Lymphoblastic Leukemia Defined by Undetectable Minimal Residual Disease: Results of an International Randomized Trial (AIEOP-BFM ALL 2000). J Clin Oncol. 2018 Jan 20;36(3):244-253. doi: 10.1200/JCO.2017.74.4946. Epub 2017 Nov 17. PMID 29148893
- [Derived] Moricke A, Zimmermann M, Valsecchi MG, Stanulla M, Biondi A, Mann G, Locatelli F, Cazzaniga G, Niggli F, Arico M, Bartram CR, Attarbaschi A, Silvestri D, Beier R, Basso G, Ratei R, Kulozik AE, Lo Nigro L, Kremens B, Greiner J, Parasole R, Harbott J, Caruso R, von Stackelberg A, Barisone E, Rossig C, Conter V, Schrappe M. Dexamethasone vs prednisone in induction treatment of pediatric ALL: results of the randomized trial AIEOP-BFM ALL 2000. Blood. 2016 Apr 28;127(17):2101-12. doi: 10.1182/blood-2015-09-670729. Epub 2016 Feb 17. PMID 26888258
- [Derived] Conter V, Valsecchi MG, Buldini B, Parasole R, Locatelli F, Colombini A, Rizzari C, Putti MC, Barisone E, Lo Nigro L, Santoro N, Ziino O, Pession A, Testi AM, Micalizzi C, Casale F, Pierani P, Cesaro S, Cellini M, Silvestri D, Cazzaniga G, Biondi A, Basso G. Early T-cell precursor acute lymphoblastic leukaemia in children treated in AIEOP centres with AIEOP-BFM protocols: a retrospective analysis. Lancet Haematol. 2016 Feb;3(2):e80-6. doi: 10.1016/S2352-3026(15)00254-9. Epub 2016 Jan 26. PMID 26853647
- [Derived] Conter V, Valsecchi MG, Parasole R, Putti MC, Locatelli F, Barisone E, Lo Nigro L, Santoro N, Arico M, Ziino O, Pession A, Testi AM, Micalizzi C, Casale F, Zecca M, Casazza G, Tamaro P, La Barba G, Notarangelo LD, Silvestri D, Colombini A, Rizzari C, Biondi A, Masera G, Basso G. Childhood high-risk acute lymphoblastic leukemia in first remission: results after chemotherapy or transplant from the AIEOP ALL 2000 study. Blood. 2014 Mar 6;123(10):1470-8. doi: 10.1182/blood-2013-10-532598. Epub 2014 Jan 10. PMID 24415536
- [Derived] Schrappe M, Valsecchi MG, Bartram CR, Schrauder A, Panzer-Grumayer R, Moricke A, Parasole R, Zimmermann M, Dworzak M, Buldini B, Reiter A, Basso G, Klingebiel T, Messina C, Ratei R, Cazzaniga G, Koehler R, Locatelli F, Schafer BW, Arico M, Welte K, van Dongen JJ, Gadner H, Biondi A, Conter V. Late MRD response determines relapse risk overall and in subsets of childhood T-cell ALL: results of the AIEOP-BFM-ALL 2000 study. Blood. 2011 Aug 25;118(8):2077-84. doi: 10.1182/blood-2011-03-338707. Epub 2011 Jun 30. PMID 21719599
- [Derived] Conter V, Bartram CR, Valsecchi MG, Schrauder A, Panzer-Grumayer R, Moricke A, Arico M, Zimmermann M, Mann G, De Rossi G, Stanulla M, Locatelli F, Basso G, Niggli F, Barisone E, Henze G, Ludwig WD, Haas OA, Cazzaniga G, Koehler R, Silvestri D, Bradtke J, Parasole R, Beier R, van Dongen JJ, Biondi A, Schrappe M. Molecular response to treatment redefines all prognostic factors in children and adolescents with B-cell precursor acute lymphoblastic leukemia: results in 3184 patients of the AIEOP-BFM ALL 2000 study. Blood. 2010 Apr 22;115(16):3206-14. doi: 10.1182/blood-2009-10-248146. Epub 2010 Feb 12. PMID 20154213